CLINICAL TRIAL: NCT01666574
Title: The Effect of Oat Based Breakfast Cereals on Satiety and Food Intake.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: PepsiCo Global R&D (Industry); Quaker Oats Company (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 12029 (Period 2)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Food Intake; Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test cereal 1, Oat-based (Experimental): The purpose of this arm is to determine if a breakfast containing 250 kcal of Oat based cereal will cause people to eat less at lunch.
  Interventions: Other: Test cereal 1, Oat-based; Other: Test Cereal 2, Oat based
- Test Cereal 2, Oat based (Experimental): The purpose of this arm is to determine if a breakfast containing 250 kcal of Oat based ready-to-eat cereal will cause people to eat less at lunch.
  Interventions: Other: Test cereal 1, Oat-based; Other: Test Cereal 2, Oat based

INTERVENTIONS:
Other: Test cereal 1, Oat-based — The study design is a lunch that will be presented 4 hours after the start of breakfast. Subjects will be asked to eat until satisfied and food intake will will be measured. The effect on hunger and satiety will be measured using visual analog scales before breakfast and at 30, 60, 120, 180, and 240 minutes following consumption.
Other: Test Cereal 2, Oat based — The study design is a two visit trial with each subject randomly receiving one of the cereals at each visit separated by at least a week. A lunch will be presented 4 hours after the start of breakfast. Subjects will be asked to eat until satisfied and food intake will be measured. The effect on hunger and satiety will be measured using visual analog scales before breakfast and at 30, 60, 120, 180, and 240 minutes following consumption.

SUMMARY:
This study is to determine if two breakfasts of equivalent calories, an oat based breakfast cereal or a ready-to-eat cereal, provide the same satiety benefits. The study will also determine if the two calorically equivalent oat-based breakfast cereals give different caloric intakes at a lunch meal that participants will eat to their satisfaction.

DETAILED DESCRIPTION:
The Second trial (Period 2): An additional 48 healthy men and women 18 years of age or older will be enrolled to investigate the satiety and food intake at lunch after a breakfast consisting of one of two randomly assigned oat-based cereals and milk breakfast. Visual analogue scales of hunger and satiety will be completed before breakfast and at, 30, 60, 120, 180, and 240 minutes following consumption. Subjects will be asked to eat Lunch until satisfied. The subjects will have the two breakfasts in a balanced and random order and the two meal tests will be separated by at least a week.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and are healthy.
* Taking no regular medications other than birth control or hormone replacement therapy.
* Are willing to use an effective method of birth control if you are capable of bearing children. Acceptable methods include abstinence, barrier methods, intrauterine devices, and hormonal methods of contraception.

Exclusion Criteria:

* Are a woman who is pregnant or nursing a baby.
* Have gained or lost 8.8 pounds or more in the last 3 months.
* Have diabetes or a fasting blood sugar over 126 mg/dL.
* Have a score of 14 or greater on the restraint scale of the 3-factor eating questionnaire (a questionnaire which will be given to you by the study staff).
* Are allergic to oats, lactose-free milk, Honey Nut Cheerios or oatmeal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Satiety Impact | Baseline to 2 days
  Breakfast containing 250 kcal of Oat-based breakfast cereal will cause people to eat less at lunch compared to a breakfast containing 250 kcal of the ready-to-eat oat-based breakfast cereal. Area under the curve (AUC) of appetite and satiety.

SECONDARY OUTCOMES:
Impact on food intake at lunch | Baseline to 2 days
  You will fill out a visual analog scales at 30, 60, 120, 180, and 240 minutes following the start of the breakfast meal each day.
  Four hours after the start of breakfast, you will be presented with a lunch and will be asked to eat to your satisfaction over 20 minutes. You will be asked how you are feeling periodically throughout the test. Area under the curve for subjective energy measures

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States